CLINICAL TRIAL: NCT06599671
Title: Effectiveness of Transvaginal Niche Resection Versus Expectant Management in Patients with Secondary Infertility and a Large Uterine Caesarean Scar Defect (niche), a Randomised Controlled Trial
Brief Title: Effectiveness of Transvaginal Niche Resection Versus Expectant Management in Patients with Secondary Infertility and a Large Uterine Caesarean Scar Defect
Acronym: TVARES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-10
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Caesarean Scar Defect
Keywords: caesarean scar defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transvaginal niche resection (Experimental): The patients assigned to the intervention group will undergo a procedure under general anaesthesia in lithotomy position.
  Interventions: Procedure: Transvaginal niche resection
- Standard of care (No Intervention): The patients assigned to the control group will receive usual care at least 9 months which means no additional surgical intervention during this period.

INTERVENTIONS:
Procedure: Transvaginal niche resection — In short: the bladder was carefully dissected away from the uterus towards the abdominal cavity to open the vesicovaginal space and reach the peritoneum. The fingers on the anterior wall isthmus could touch the obvious scar-like defect. The weak scar tissue then thoroughly was removed.
  Arms: Transvaginal niche resection

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of transvaginal niche resection in improving pregnancy outcomes of a large uterine caesarean scar defect (niche) with secondary infertility. The main questions it aims to answer are:

1. Does transvaginal niche resection improve pregnancy outcomes of a large uterine caesarean scar defect (niche) with secondary infertility?
2. What medical problems do participants have when taking transvaginal niche resection?

Researchers will compare transvaginal niche resection to expectant management (without any additional surgical intervention) to see if transvaginal niche resection works to improve pregnancy outcomes of a large uterine caesarean scar defect (niche) with secondary infertility.

Participants will:

1. Undergo a procedure (transvaginal niche resection) within 2 week after randomization in the intervention group. Women were advised to use contraception in the first 6 months following niche resection to allow uterine healing prior to subsequent pregnancy.
2. Receive usual care at least 9 months which means no additional surgical intervention during this period in the control group. Patients are allowed to become pregnant and to receive fertility therapies if indicated. Any member of the control group who has not become pregnant after 9 months will be given the opportunity to undergo a transvaginal niche resection.
3. Receive a standardized magnetic resonance imaging (MRI) evaluation of the niches. Niches will be evaluated at baseline in all groups and at 3 months after surgery.
4. Be contacted by telephone at 6, 9 and 15 months to assess the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. It was diagnosed by MRI as a large niche (defined as niche with a depth of >50% of the myometrial thickness and a residual myometrial thickness (RMT) ≤3mm);
2. Infertility secondary to niche (the inability to conceive within 12 months of unprotected intercourse or repeated failed IVF);
3. Fertility requirements;
4. Signed informed consent.

Exclusion Criteria:

1. Age below 18 years or over 49 years;
2. Contraindications for intraspinal or general anaesthesia;
3. A (suspected) malignancy or combined benign lesions requiring hysterectomy;
4. Atypical endometrial cells or cervical dysplasia;
5. Uterine or cervical polyps;
6. Submucosal fibroids;
7. Hydrosalpinx.

Ages: 19 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Total follow-up will extend to 15 months after randomization.
  Live birth is defined as a live born neonate beyond 24 weeks of gestation.

IPD SHARING:
Plan to Share IPD: No